CLINICAL TRIAL: NCT04891783
Title: Investigating Atherosclerosis In Seronegative Spondyloarthropathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Salma Mohamed Shabaan, assistant lecturer, Sohag University
Other Study IDs: Soh-Med-21-05-11
Record Dates: First submitted 2021-05-17; First posted 2021-05-18 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: In Seronegative Spondyloarthropathy
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 50 patients diagnosed as AS: 50 patients diagnosed as AS according to 1984 modified New York criteria of AS .including radiographic and non-radiographic AS according to ASAS criteria these patients will undergo carotid ultrasound examination
  Interventions: Device: ultrasonography
- 30 patients with psoriatic arthritis: 30 patients with psoriatic arthritis who will be diagnosed according to the Classification Criteria of Psoriatic Arthritis (CASPAR) study these patients will undergo carotid ultrasound examination
  Interventions: Device: ultrasonography
- 40 healthy controls: healthy controls will undergo carotid ultrasound examination
  Interventions: Device: ultrasonography

INTERVENTIONS:
Device: ultrasonography — The Carotid US examination will be performed by a radiologist, according to the same protocol in the different participating hospitals. It will include the measurement of cIMT in the common carotid artery and the detection of focal plaques in the extracranial carotid tree following the Mannheimconsensus[26]. Plaque is defined as a focal protrusion in the lumen at least cIMT>1.5 mm, protrusion at least 50% greater than the surrounding cIMT, or arterial lumen encroaching >0.5 mm [26]. The cIMT will be determined as the average of three measurements in each common carotid artery. The final cIMT is the largest average cIMT (left or right). Patients with carotid plaques will be considered as having very high CV .
  Other Names: MRI

SUMMARY:
The association between inflammation and atherosclerosis is widely known. An increase in morbidity and mortality due to cardiovascular (CV) disease in inflammatory rheumatic diseases has been proved [1-4]. Rheumatoid arthritis (RA) has the greatest CV impact. Scientific societies and expert groups have developed recommendations for preventing cardiovascular risk in these patients [5, 6]. It has also been observed an increased CV risk and greater morbidity in other inflammatory rheumatic diseases such as Ankylosing Spondylitis (AS), psoriatic arthritis (PsA), and inflammatory bowel disease(IBD) [1, 7n, 8].

Ankylosing spondylitis (AS) is a systemic inflammatory disorder of unknown etiology that mainly involves the axial skeleton causing the spine, sacroiliac joints arthritis, and peripheral joints arthritis. Its peak age of onset is between 20-30 years affecting young males with the involvement of extra-articular structures such as eyes, kidneys, heart, lung, vessels, and nerves [9,10]. Aortitis and aortic regurgitation are cardiovascular complications associated with AS. AS is associated with up to 50% mortality rates and cardiovascular diseases are the main causes of these high mortality rates[10,11].

DETAILED DESCRIPTION:
The association between inflammation and atherosclerosis is widely known. An increase in morbidity and mortality due to cardiovascular (CV) disease in inflammatory rheumatic diseases has been proved . Rheumatoid arthritis (RA) has the greatest CV impact. Scientific societies and expert groups have developed recommendations for preventing cardiovascular risk in these patients . It has also been observed an increased CV risk and greater morbidity in other inflammatory rheumatic diseases such as Ankylosing Spondylitis (AS), psoriatic arthritis (PsA), and inflammatory bowel disease(IBD).

Ankylosing spondylitis (AS) is a systemic inflammatory disorder of unknown etiology that mainly involves the axial skeleton causing the spine, sacroiliac joints arthritis, and peripheral joints arthritis. Its peak age of onset is between 20-30 years affecting young males with the involvement of extra-articular structures such as eyes, kidneys, heart, lung, vessels, and nerves [9,10]. Aortitis and aortic regurgitation are cardiovascular complications associated with AS. AS is associated with up to 50% mortality rates and cardiovascular diseases are the main causes of these high mortality rates.

The psoriatic disease concept includes psoriatic arthritis (PsA). PsA is a chronic inflammatory skeletal disease associated with psoriasis. PsA has heterogeneous clinical manifestations with some forms linked to the spondyloarthritis(SpA) concept. A strong relationship of PsA with SpA is clearly supported by shared clinical, genetic, and radiographic characteristics.

CV comorbidities are critically important in this patient population because they may directly contribute to increased mortality seen in patients PsA.

Sustained chronic systemic inflammation predisposes to atherosclerosis as it is accompanied by elevated levels of serum C-reactive protein (CRP), which has proatherogenic effects. Also, hypertension, sex, and smoking are predisposing factors with chronic inflammation in atherosclerosis.3 Moreover, AS has been associated with a prevalence of metabolic syndrome including dyslipidemia and a high ratio of low-density lipoprotein (LDL) cholesterol to high-density lipoprotein (HDL) cholesterol .

SerumIrisin, asa novel hormone-like myokine that plays a pivotal role in energy expenditure and metabolic regulation, is mainly secreted by the heart, skeletal muscle, liver, kidneys, nerves

, and skin.Previous studies revealed the relationship between circulating irisin levels, endothelial dysfunctions, and subclinical atherosclerosis in non-diabetic adult patients.[18]In another recent study, it was demonstrated that serum irisin level was significantly correlated with carotid atherosclerosis in patients receiving dialysis.

As a consequence of the aforementioned considerations, the prevention of CV events has become an issue of great concern in the treatment of chronic inflammatory diseases. Primary prevention strategies designed for the general population are based on the performance of composite scores to estimate the total CV risk, thus identifying those individuals at higher risk who may benefit from active therapy. The 2019 ESC/EAS guidelines for the treatment of dyslipidemias also recommend considering the assessment of carotid plaque burden on ultrasound as a risk modifier in people with low or moderate CV risk. According to these guidelines, the presence of carotid plaques would automatically imply the reclassification of an individual as having very high CV risk [21]. This recommendation seems particularly useful for patients with inflammatory conditions, whose CV risk tends to be underestimated by composite scores because of not considering important pro-atherogenic factors related to the disease such as inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Age at disease onset above 16 yrs old
* Patients diagnosed as according to 1984 modified New York criteria of AS .including radiographic and non-radiographic AS according to ASAS crteriae[22].
* Psoriatic arthritis patients fulfilling the diagnostic criteria defined by the Classification Criteria of Psoriatic Arthritis (CASPAR[23]study and with a diagnosis confirmed by a rheumatologist

Exclusion Criteria:

* Diabetes mellitus or use of antidiabetic medication.
* Heart failure, as defined by ejection fraction <50%.
* Renal disease.
* Chronic obstructive lung disease; pulmonary hypertension; pregnancy or obesity.
* Metabolic syndrome.
* History of cardiovascular, peripheral artery disease, or cerebrovascular events.

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This study will be carried out as a case-control study on patients followed up in the Rheumatology and Rehabilitation outpatient clinic in Sohag University Hospitals, Faculty of Medicine:
  50 patients diagnosed as AS according to 1984 modified New York criteria of AS .including radiographic and non-radiographic AS according to ASAS criteria .
  30 patients with psoriatic arthritis who will be diagnosed according to the Classification Criteria of Psoriatic Arthritis (CASPAR) study And 40 healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Investigate the presence of atherosclerosis in two diseases of seronegative spondyloarthropathy ankylosing spondylitis and psoriatic arthritis patients | 2 years
  The purpose of this study is to investigate the presence of atherosclerosis based on the results of carotid ultrasound and serum irsin level in two diseases of seronegative spondyloarthropathy ankylosing spondylitis and psoriatic arthritis patients.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Shen J, Shang Q, Li EK, Leung YY, Kun EW, Kwok LW, Li M, Li TK, Zhu TY, Yu CM, Tam LS. Cumulative inflammatory burden is independently associated with increased arterial stiffness in patients with psoriatic arthritis: a prospective study. Arthritis Res Ther. 2015 Mar 17;17(1):75. doi: 10.1186/s13075-015-0570-0. PMID 25890227
- [Background] Mach F, Baigent C, Catapano AL, Koskinas KC, Casula M, Badimon L, Chapman MJ, De Backer GG, Delgado V, Ference BA, Graham IM, Halliday A, Landmesser U, Mihaylova B, Pedersen TR, Riccardi G, Richter DJ, Sabatine MS, Taskinen MR, Tokgozoglu L, Wiklund O; ESC Scientific Document Group. 2019 ESC/EAS Guidelines for the management of dyslipidaemias: lipid modification to reduce cardiovascular risk. Eur Heart J. 2020 Jan 1;41(1):111-188. doi: 10.1093/eurheartj/ehz455. No abstract available. PMID 31504418
- [Background] Taylor W, Gladman D, Helliwell P, Marchesoni A, Mease P, Mielants H; CASPAR Study Group. Classification criteria for psoriatic arthritis: development of new criteria from a large international study. Arthritis Rheum. 2006 Aug;54(8):2665-73. doi: 10.1002/art.21972. PMID 16871531